CLINICAL TRIAL: NCT03745300
Title: Comparative Evaluation Of 1.2% Atorvastatin and 1.2% Simvastatin Gel Local Drug Delivery And Redelivery In Chronic Periodontitis Subjects With Diabetes Mellitus: A Randomized Controlled Clinical Trial.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, professor and HOD, Department of periodontology, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/Ph.D/5/2016-2017H
Record Dates: First submitted 2018-11-02; First posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Chronic Periodontitis Wth Diabetes Mellitus
MeSH Terms: interventions — Atorvastatin; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GROUP 1 (Active Comparator): Scaling and root planing (SRP) followed by 1.2% atorvastatin gel local drug delivery
  Interventions: Drug: ATORVASTATIN
- GROUP 2 (Active Comparator): Scaling and root planing (SRP) followed by 1.2% simvastatin gel local drug delivery
  Interventions: Drug: SIMVASTATIN
- GROUP 3 (Placebo Comparator): Scaling and root planing (SRP) followed by placebo gel local drug delivery
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: ATORVASTATIN — Scaling and Root Planing (SRP) followed by placement of atorvastatin gel
  Other Names: ATV
  Arms: GROUP 1
Drug: SIMVASTATIN — Scaling and Root Planing (SRP) followed by placement of simvastatin gel
  Other Names: SMV
  Arms: GROUP 2
Drug: PLACEBO — Scaling and Root Planing (SRP) followed by placement of placebo gel
  Other Names: inactive drug
  Arms: GROUP 3

SUMMARY:
Statins are specific competitive inhibitors of 3-hydroxy-3-methylglutaryl coenzyme A (HMG-CoA) reductase, known for its hypolipidemic actions, possessing biologically significant anti-inflammatory and antioxidant properties, exerts anabolic effects on bone through expression of BMP - 2, have paved way in periodontal regeneration. The present study aims to evaluate and compare the efficacy of subgingivally delivered 1.2% Atorvastatin (ATV) and 1.2% Simvastatin (SMV) gel local drug delivery and redelivery systems as an adjunct to scaling and root planning (SRP) in chronic periodontitis (CP) subjects with diabetes mellitus(DM).

DETAILED DESCRIPTION:
Statins are specific competitive inhibitors of 3-hydroxy-3-methylglutaryl coenzyme A (HMG-CoA) reductase, known for its hypolipidemic actions, possessing biologically significant anti-inflammatory and antioxidant properties, exerts anabolic effects on bone through expression of BMP - 2, have paved way in periodontal regeneration. The present study aims to evaluate and compare the efficacy of subgingivally delivered 1.2% Atorvastatin (ATV) and 1.2% Simvastatin (SMV) gel local drug delivery and redelivery systems as an adjunct to scaling and root planning (SRP) in chronic periodontitis (CP) subjects with diabetes mellitus(DM). 120 subjects with intrabony defects were divided into three groups;group 1- SRP plus 1.2% ATV ; group 2- SRP PLUS 1.2% SMV; and group 3- SRP plus placebo gel. Clinical and radiographic measurements were taken at baseline, at 6 months and respective gels were redelivered subgingivally in respective groups . Measurements were repeated again at 3 months i.e. 9 months from baseline.

ELIGIBILITY:
Inclusion Criteria:

* well controlled type 2 diabetes mellitus patients classified based on criteria given by American diabetes association with CP with PD≥5mm and CAL ≥3mm and presence of IBD ≥ 3 mm (distance between alveolar crest and base of the defect on an intraoral periapical radiograph [IOPAR] after phase I therapy

Exclusion Criteria:

* 1)patients with known allergy to statins; 2) Patients with systemic conditions / medications known to affect the periodontal status; 3) aggressive and refractory periodontitis 4) Hematological disorders 5) pregnancy/lactation; and 6) Smoking and tobacco use in any form 7) Immunocompromised individuals.8). patients with poor plaque control. 9). non vital teeth, carious teeth warranting restorations, third molars and mobility of at least grade II were excluded.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
change in defect depth | 6 and 9 months
  assessed in percentage

SECONDARY OUTCOMES:
change in probing depth (PD) | baseline, 6 and 9 months
change in Clinical Attachment Level (CAL) | baseline, 6 and 9 months
CHANGE IN Plaque Index (PI) | baseline, 6 and 9 months
change in modified Sulcus Bleding Index (mSBI) | baseline, 6 and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Avani R Pradeep, MDS, Principal Investigator — GDCRI, Bangalore, INDIA
Locations (1):
- Department of Periodontics, GDCRI Bangalore, Bangalore, Karnataka, India